CLINICAL TRIAL: NCT01256021
Title: Multi-center, Single Arm, Open-label, Phase IV Clinical Trial to Evaluate the Safety and Efficacy of MEDITOXIN® in Children With Cerebral Palsy
Brief Title: The Efficacy and Safety of MEDITOXIN® in Children With Cerebral Palsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT_PRT_CP02
Record Dates: First submitted 2010-12-06; First posted 2010-12-08 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Muscle Spasticity
MeSH Terms: conditions — Muscle Spasticity | interventions — Botulinum Toxins, Type A; 3-deoxyglycero-galacto-nonulosonic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Group 1 (Experimental): Meditoxin
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A — 1 time, gastrocnemius muscles injection, dose of 4U/kg body weight in patients with hemiplegia, dose of 6U/kg body weight in patients with diplegia, Maximum dosage 200U
  Other Names: Neuronox®, Siax®

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Meditoxin® in the treatment of children with cerebral palsy.

DETAILED DESCRIPTION:
The allocated subject is injected Meditoxin® 4U/kg body weight(for patients with hemiplegia) or 6U/kg body weight(for patients with diplegia)in the affected gastrocnemius muscle for the treatment of patients who suffer Equinus Foot Deformity with pediatric cerebral palsy due to spasticity.

The efficacy and safety are evaluated for 12weeks through 3 follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged between 2 and 18 years with diagnosis of spastic cerebral palsy
* Patients with toe-walking due to peroneal muscle spasticity (patients with equinus foot deformity due to spasticity)
* Patients who voluntarily consent to participate in this study and whose legally acceptable representative has signed the informed consent form (if the patient is able to write, his/her signature should be also obtained).

Exclusion Criteria:

* Patients who had previously received botulinum toxin within 3 months prior to the study entry
* Patients with known hypersensitivity to botulinum toxin
* Patients who requires legs, feet or ankle surgery at present
* Patients with severe athetoid movement
* Patients who is participating in other investigational study at present
* Patients, by the investigator's discretion, who are not suitable for this study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 212 (Actual)
Dates: Start 2010-08; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in MAS score from baseline to week 4 | 4 weeks
  The investigator assessed MAS score using a 5-point scale (0, 1, 1+, 2, 3, and 4; 0=No increase in muscle tone to 4=Affected part[s] rigid in flexion or extension) The "+1" (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder [less than half] of ROM [range of motion]) of MAS score is regarded as score 2

SECONDARY OUTCOMES:
Mean change from baseline in MAS score from baseline to week 12 | 12 weeks
  The investigator assessed MAS score using a 5-point scale (0, 1, 1+, 2, 3, and 4; 0=No increase in muscle tone to 4=Affected part[s] rigid in flexion or extension) The "+1" (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder [less than half] of ROM [range of motion]) of MAS score is regarded as score 2
Mean change from baseline in PROM(Passive Range of Motion of ankle) at ankle dorsiflexion from baseline to week 4, 12 | 4, 12 Weeks
Mean change from baseline in VAS(Visual Analogue Scale)assessed by caregiver/patient from baseline to week4 | 4, 12 weeks
  Individual goals of treatment were chosen one among pain, ease of care, standing, walking. The VAS used in this study is a straight 10cm horizontal line with anchor points of very satisfied (score 0)and very dissatisfied (score 10).
Improvement in Global Assessment assessed by caregiver/patient | 4, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eun S Park, Ph D, Principal Investigator — Severance Hospital
Locations (4):
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National Universtiy Hospital, Seoul
  - Asan Medical Center, Seoul
  - Yonsei University Severance Hospital, Seoul